CLINICAL TRIAL: NCT02379546
Title: The Effect of Anaesthesia Depth on Oculo-cardiac Reflex in Strabismus Surgery
Brief Title: The Effect of Anaesthesia Depth on Oculo-cardiac Reflex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Tuğba Karaman, assistant professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GaziosmanpashaU-2
Record Dates: First submitted 2015-02-17; First posted 2015-03-05 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Strabismus; Anesthesia, General
Keywords: reflex, oculocardiac; monitoring, intraoperative
MeSH Terms: conditions — Strabismus | interventions — Desflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BIS<50 (Experimental): Anaesthesia will be maintained with desflurane in a 50% O2-Air mixture by titrating the concentration according to the Bispectral index monitoring to keep the Bispectral index values below 50.
  Interventions: Drug: Desflurane; Device: Bispectral index monitoring
- BIS≥50 (Active Comparator): Anaesthesia will be maintained with desflurane in a 50% O2-Air mixture by titrating the concentration according to the Bispectral index monitoring to keep the Bispectral index values above 50.
  Interventions: Drug: Desflurane; Device: Bispectral index monitoring

INTERVENTIONS:
Drug: Desflurane — Desflurane will be used to maintain the anesthesia and the dose of desflurane will be adjusted according to the Bispectral İndex Monitoring
Device: Bispectral index monitoring — Bispectral index monitoring (BIS XP, A-2000, VERSİON 3.31, Aspect Medical Systems, Newton, Mass, USA)will be used to determine the depth of anesthesia
  Other Names: BIS

SUMMARY:
This study was designed to determine the effect of the depth of anesthesia on the oculocardiac reflex (OCR) during pediatric strabismus surgery.

DETAILED DESCRIPTION:
The oculo-cardiac reflex (OCR) is a trigeminovagal reflex which is started by the stimulus on the extra-ocular muscle and may lead to serious bradycardia or arrhythmia in the patients during strabismus surgery. It is presumed that the depth of anesthesia is one of the influencing factor on the OCR. But the clinical trials which are evaluating the relationship between the anesthesia depth and OCR are scarce. The main objective of this study is to determine the impact of the depth of anaesthesia that is adjusted with the bispectral index (BIS) monitor on the incidence of OCR in pediatric patients undergoing strabismus surgery.

ELIGIBILITY:
Inclusion Criteria:

* physical status ASA (American Society of Anesthesiologists) I
* scheduled for elective strabismus surgery under general anesthesia
* aged between 3-16 years

Exclusion Criteria:

* have a neurological or cardiovascular disease
* receiving antiepileptic or another medications known to affect EEG or ECG

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2013-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The effect of the anaesthesia depth on the incidence of oculocardiac reflex | during the traction of the extra-ocular muscle in the strabismus surgery

SECONDARY OUTCOMES:
The incidence of the oculocardiac reflex depending the type of operated extra-ocular muscle during the strabismus surgery | during the traction of the extra-ocular muscle in the strabismus surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Karaman, Principal Investigator — GOU
Locations (1):
- Tuğba Karaman, Tokat Province, Merkez, Turkey (Türkiye)